CLINICAL TRIAL: NCT05436067
Title: Evaluation of an App for Individualized Vestibular Rehabilitation for Elderly With Self-Management and Gaming Elements
Brief Title: Individualized Vestibular Rehabilitation for Elderly With Self-Management and Gaming Elements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CFD Research Corporation (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00148324; 5R44DC017408-03 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-28 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Disorder; Balance; Distorted; Vestibular Diseases
Keywords: balance; telehealth; physical therapy; mobile application; serious gaming; rehabilitation; vestibular; dizziness
MeSH Terms: conditions — Vestibular Diseases; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trials with Vestibular Rehabilitation App (Experimental): All participants underwent the same experiment. They will performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
  This arm describes the results of the trials where exercises were performed with the Vestibular Rehabilitation App.
  Interventions: Device: Vestibular rehabilitation app
- Trials without Vestibular Rehabilitation App (Experimental): All participants underwent the same experiment. They will performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
  This arm describes the results of the trials where exercises were performed without the Vestibular Rehabilitation App.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Device: Vestibular rehabilitation app — Delivery of vestibular rehabilitation through an app on a tablet or other portable device. The app takes patients through their rehabilitation session that has been prescribed by a clinician. Exercises are presented in the forms of games that are controlled by head or torso motion via a motion sensor that is placed on that body part. Data on the motion of the patient are calculated from sensor data and sent over the cloud for the clinician to access remotely.
  Arms: Trials with Vestibular Rehabilitation App
Other: Traditional Physical Therapy — Delivery of vestibular rehabilitation through traditional physical therapy.
  Arms: Trials without Vestibular Rehabilitation App

SUMMARY:
The aim of this study is to test whether when using the Vestibular Rehabilitation App older patients perform rehabilitation in a similar manner as when directly instructed by a clinician. A secondary goal is to evaluate usability and enjoyment of the app.

DETAILED DESCRIPTION:
The main aim of this study is to test the prototype Vestibular Rehabilitation App (that has been specifically developed for this study) in the lab setting to evaluate if patients perform exercises with the app in a similar manner as when performing exercises in the traditional manner without the app. Errors in exercise performance identified by the app will be compared to those identified by a physical therapist. A secondary aim is to get feedback on enjoyment and ease of use of the Vestibular Rehabilitation App.

ELIGIBILITY:
Inclusion Criteria:

* aged between 60 and 75
* Presence of dizziness due to a central or peripheral vestibular disorder

Exclusion Criteria:

* Presence of neurological disease such as stroke, multiple sclerosis, Parkinson's
* History of recent lower extremity surgery or severe pain in legs

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulien Roos, PhD, Principal Investigator — CFD Research Corporation
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
All resources developed for this project will be presented at conferences and published in the literature where possible. Whenever possible the investigators will include supplemental data (de-identified) in the online versions of their publications to most fully disseminate our results. Also, resources and de-identified data will be made available, whenever possible and appropriate, to qualified persons upon request.
Time Frame: Data will be available upon request after they have been published
Access Criteria: Upon request

REFERENCES:
- [Background] DSilva LJ, Skop KM, Pickle NT, Marschner K, Zehnbauer TP, Rossi M, Roos PE. Use of Stakeholder Feedback to Develop an App for Vestibular Rehabilitation-Input From Clinicians and Healthy Older Adults. Front Neurol. 2022 Feb 24;13:836571. doi: 10.3389/fneur.2022.836571. eCollection 2022. PMID 35280295
- [Background] Davis, F. D. Perceived Usefulness, Perceived Ease of Use, and User Acceptance of Information Technology. MIS Quarterly. 1989; 13(3): 319-340.
- [Background] Chin, J.P., Diehl, V.A., and Norman, K.L. Development of a tool measuring user satisfaction of the human-computer interface. CHI '88: Proceedings of the SIGCHI Conference on Human Factors in Computing Systems. 1988; 213-218.
- [Background] van Het Reve E, Silveira P, Daniel F, Casati F, de Bruin ED. Tablet-based strength-balance training to motivate and improve adherence to exercise in independently living older people: part 2 of a phase II preclinical exploratory trial. J Med Internet Res. 2014 Jun 25;16(6):e159. doi: 10.2196/jmir.3055. PMID 24966165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants were recruited and participated in this study.
Groups:
- Older Adults With Dizziness: All participants underwent the same experiment. They performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
Period: Overall Study
Arm/Group | Older Adults With Dizziness
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All participants underwent the same experiment. They will performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
  In the rest of the reporting the overall study population is presented in two different arms, "Trials with Vestibular Rehabilitation App" and "Trials without Vestibular Rehabilitation App". These are the same participants and all participated in both arms.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.65 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Perceived Usefulness
Description: The ease of use of information technology questionnaire is used to rate usefulness and perceived ease of use of the Vestibular Rehabilitation app. These are rated on a scale of 1-7, with 1 being the most positive response, 4 being a neutral response and 7 being the most negative response.
Time Frame: Immediately after the testing
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Older Adults With Dizziness: Clinical trial only has one arm or participant group. All participants undergo the same experiment. They will perform exercises with the Vestibular Rehabilitation App as well as without the App. The order is randomized.
  Vestibular rehabilitation app: Delivery of vestibular rehabilitation through an app on a tablet or other portable device. The app takes patients through their rehabilitation session that has been prescribed by a clinician. Exercises are presented in the forms of games that are controlled by head or torso motion via a motion sensor that is placed on that body part. Data on the motion of the patient are calculated from sensor data and sent over the cloud for the clinician to access remotely.
Arm/Group | Older Adults With Dizziness
Number analyzed (Participants) | 40
units on a scale | 1.99 (1.00)

2. Primary Outcome: User Interface Satisfaction Questionnaire Outcomes
Description: The questionnaire for user interface satisfaction (QUIS) is used to rate the Vestibular Rehabilitation app on use of its software and screen. These are rated on a scale of 0-9, with 9 being the most positive response and 0 being the most negative response.
Time Frame: Immediately after the testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Adults With Dizziness
Number analyzed (Participants) | 40
units on a scale | 7.59 (1.70)

3. Primary Outcome: Use Intention, Motivation and Enjoyment
Description: A questionnaire on use intention, motivation, and enjoyment is used to rate the Vestibular Rehabilitation app on the use intention, motivation and enjoyment of the app. These are rated on a scale of 1-7, with 1 being the most positive response, 4 being a neutral response and 7 being the most negative response.
Time Frame: Immediately after the testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Adults With Dizziness
Number analyzed (Participants) | 40
units on a scale | 1.90 (1.13)

4. Primary Outcome: Change in Head Angle With the App
Description: The IMU sensor data collected during the exercise performance with and without the Vestibular Rehabilitation App (collected in the same lab visit on the same group of participants) were analyzed to calculate peak head angles. These were analyzed to identify differences for the conditions with and without the Vestibular Rehabilitation App.
Time Frame: During the testing with the app and during the testing without the app (up to 90 minutes)
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Trials With the Vestibular Rehabilitation App: All participants underwent the same experiment. They performed exercises with the Vestibular Rehabilitation App as well as without the App and this occurred in the same lab visit. The order is randomized. these different trials with and without the app are presented as separate arms. This arms concerns the trials with the Vestibular Rehabilitation App.
- Trials Without the Vestibular Rehabilitation App: All participants underwent the same experiment. They performed exercises with the Vestibular Rehabilitation App as well as without the App and this occurred in the same lab visit. The order is randomized. these different trials with and without the app are presented as separate arms. This arms concerns the trials without the Vestibular Rehabilitation App.
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without the Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 40
degrees
  Peak pitch angle - left | 13.2 (6.9) | 22.0 (8.3)
  Peak pitch angle - right | 13.8 (7.8) | 21.4 (8.2)
  Peak yaw angle - flexion | 13.6 (6.0) | 16.0 (13.2)
  Peak yaw angle - extension | 14.7 (5.7) | 16.5 (10.8)
Statistical Analysis 1: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p < 0.001, paired t-test — Difference in head angle pitch - left between the arms
Statistical Analysis 2: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p < 0.001, paired t-test — Difference in head angle pitch - right between the arms
Statistical Analysis 3: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p = 0.042, paired t-test — Difference in head angle yaw - extension between the arms
Statistical Analysis 4: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p = 0.111, paired t-test — Difference in head angle yaw - flexion between the arms

5. Primary Outcome: Change in Range of Motion With the App
Description: The IMU sensor data collected during the exercise performance with and without the Vestibular Rehabilitation App (collected in the same lab visit on the same group of participants) were analyzed to calculate head range of motion values. These were analyzed to identify differences for the conditions with and without the Vestibular Rehabilitation App
Time Frame: During the testing with the app and during the testing without the app (up to 90 minutes)
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Trials Without Vestibular Rehabilitation App: All participants underwent the same experiment. They performed exercises with the Vestibular Rehabilitation App as well as without the App and this occurred in the same lab visit. The order is randomized. these different trials with and without the app are presented as separate arms. This arms concerns the trials without the Vestibular Rehabilitation App.
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 40
degrees
  Range of motion - yaw | 14.1 (5.3) | 16.6 (7.0)
  Range of motion - pitch | 13.6 (7.0) | 22.9 (9.7)
Statistical Analysis 1: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p = 0.023, paired t-test — Difference in pitch range of motion between the arms
Statistical Analysis 2: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p < 0.001, paired t-test

6. Primary Outcome: Change in Head Motion Frequency With the App
Description: The IMU sensor data collected during the exercise performance with and without the Vestibular Rehabilitation App (collected in the same lab visit on the same group of participants) were analyzed to calculate frequency of head motion. These were analyzed to identify differences for the conditions (arms) with and without the Vestibular Rehabilitation App
Time Frame: During the testing with the app and during the testing without the app (up to 90 minutes)
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without the Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 40
Hz
  Pitch frequency | 0.93 (0.1) | 0.93 (0.27)
  Yaw frequency | 0.93 (0.13) | 0.85 (0.27)
Statistical Analysis 1: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p = 0.057, paired t-test — Difference in pitch velocity between the arms
Statistical Analysis 2: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; This statistical analysis tests the difference between the different arms (with and without app) using a paired t-test; Test type: Other; p = 0.003, paired t-test — Difference in yaw velocity between the arms

7. Primary Outcome: Change in Balance Outcome With the App - Weight Shift Exercise
Description: The IMU sensor data collected during the exercise performance with and without the Vestibular Rehabilitation App (collected in the same lab visit on the same group of participants) were analyzed to calculate range of motion in different directions during the weight shift balance exercise (in degrees). These were analyzed to identify differences for the conditions with and without the Vestibular Rehabilitation App
Time Frame: During the testing with the app and during the testing without the app (up to 90 minutes)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without the Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 40
degrees
  Weight shift exercise - mediolateral range of motion | 8.7 (3.5) | 7.2 (3.5)
  Weight shift exercise - anterioposterior range of motion | 4.5 (1.6) | 3.7 (1.7)
  Single leg balance - range of motion | 8.8 (4.8) | 11.0 (6.8)
Statistical Analysis 1: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; Test type: Other; p = 0.035, paired t-test — Weight shift exercise - mediolateral range of motion
Statistical Analysis 2: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; Test type: Other; p = 0.006, paired t-test — Weight shift balance exercise anteroposterior range of motion
Statistical Analysis 3: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; Test type: Other; p = 0.024, paired t-test — Single leg balance range of motion
Statistical Analysis 4: Comparison: Trials With the Vestibular Rehabilitation App vs Trials Without the Vestibular Rehabilitation App; Test type: Other; p = 0.257, Shapiro Wilcoxon test — Single leg balance fluency; Data was not normally distributed

8. Primary Outcome: Change in Head Angle With Feedback
Description: The IMU sensor data collected during the exercise performance with the Vestibular Rehabilitation App will be analyzed to calculate peak head angles. Averages will be calculated for time windows before and after feedback on exercise performance is given. This will be analyzed to identify differences before and after feedback has been given.
Time Frame: During the testing with the app (up to 45 minutes)
Population: No participants were analyzed because too few participants received feedback during the trials. For participants that did receive feedback the time window before and after the feedback varied widely, since feedback could be provided at any point in time during the trial. Due to these inconsistencies it was decided not to perform any statistically analyses on these data or to extract and analyze these data.
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change in Range of Motion With Feedback
Description: The IMU sensor data collected during the exercise performance with the Vestibular Rehabilitation App will be analyzed to calculate range of motion values. Averages will be calculated for time windows before and after feedback on exercise performance is given. This will be analyzed to identify differences before and after feedback has been given.
Time Frame: During the intervention with the app (up to 45 minutes)
Population: No data were collected on this. The feedback was mostly provided at the start of the trial and because of this there was no time window before the feedback, which would be required to calculate the change.
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change in Angular Velocity With Feedback
Description: The IMU sensor data collected during the exercise performance with the Vestibular Rehabilitation App will be analyzed to calculate angular velocity values . Averages will be calculated for time windows before and after feedback on exercise performance is given. This will be analyzed to identify differences before and after feedback has been given.
Time Frame: During the intervention with the app (up to 45 minutes)
Population: as for outcome 9
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Change in Balance Outcome With Feedback
Description: The IMU sensor data collected during the exercise performance with the Vestibular Rehabilitation App will be analyzed to calculate balance measures (jerk). Averages will be calculated for time windows before and after feedback on exercise performance is given. This will be analyzed to identify differences before and after feedback has been given.
Time Frame: During the intervention with the app (up to 45 minutes)
Population: as for outcome 9
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Error Identification Differences
Description: The exercise errors that are identified by the Vestibular Rehabilitation App and those identified by the physical therapist will be compared.
Time Frame: During the intervention with the app (up to 45 minutes)
Population: as for outcome 9
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Open Ended Feedback
Description: Participants will be asked for open ended feedback after the testing with and without the Vestibular Rehabilitation App. Discussions will be guided with questions. The questions were as follows: 1) Describe your overall experience as you used the app today?; 2) Explain the positive features of the app as you did your exercises?; 3) Describe the negative features of the app as you did your exercises today?; 4) What changes would you like to see in the app to support you as you do your exercises?; 5) Do you see any barriers to using the app while doing your exercises at home?
Time Frame: Immediately after the intervention
Population: The open ended questions referred to the use of the Vestibular Rehabilitation App and were therefore only filled out with regards to the arm "Trials with the Vestibular Rehabilitation App"
Measure: Count of Participants; unit: Participants
Groups:
- Trials With Vestibular Rehabilitation App: All participants underwent the same experiment. They will performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
  This arm describes the results of the trials where exercises were performed with the Vestibular Rehabilitation App.
  Vestibular rehabilitation app: Delivery of vestibular rehabilitation through an app on a tablet or other portable device. The app takes patients through their rehabilitation session that has been prescribed by a clinician. Exercises are presented in the forms of games that are controlled by head or torso motion via a motion sensor that is placed on that body part. Data on the motion of the patient are calculated from sensor data and sent over the cloud for the clinician to access remotely.
- Trials Without Vestibular Rehabilitation App: All participants underwent the same experiment. They will performed exercises with the Vestibular Rehabilitation App as well as without the App. The order was randomized.
  This arm describes the results of the trials where exercises were performed without the Vestibular Rehabilitation App.
  Traditional Physical Therapy: Delivery of vestibular rehabilitation through traditional physical therapy.
Arm/Group | Trials With Vestibular Rehabilitation App | Trials Without Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 0
Participants
  Overall experience - not challenging | 1 | 0
  Overall experience - positive or fun | 30 | 0
  Overall experience - easy or easy to understand | 11 | 0
  Overall experience - engaging or interesting | 6 | 0
  Overall experience - motivating | 9 | 0
  Overall experience - difficult | 1 | 0
  Overall experience - seems geared toward more younger adults | 5 | 0
  Overall experience - not motivating | 2 | 0
  Overall experience - challenging (in a positive way) | 2 | 0
  Overall experience - reduced anxiety | 1 | 0
  Positive features - fun | 5 | 0
  Positive features - motivating | 5 | 0
  Positive features - provides feedback | 3 | 0
  Positive features - challenging | 1 | 0
  Positive features - colorful | 2 | 0
  Positive features - easy to use | 4 | 0
  Positive features - helpful | 2 | 0
  Positive feedback - seeing progress or accomplishments | 2 | 0
  Positive feedback - liked scoring or rewards | 2 | 0
  Positive feedback - liked the gaming element | 2 | 0
  Negative features - none noted | 19 | 0
  Negative features - feedback interrupted flow | 2 | 0
  Negative feedback - redundant instructions | 2 | 0
  Negative feedback - frustration with motion control | 6 | 0
  Negative feedback - learning curve | 1 | 0
  Negative feedback - transition from weight shifting to balance games was challenging | 1 | 0
  Negative feedback - juvenile theme | 5 | 0
  Negative feedback - longer setup than traditional therapy | 1 | 0
  Negative feedback - may get boring after a while | 1 | 0
  Negative feedback - colors may be hard with color blindness in some games | 1 | 0
  Would like - motion sensing improvement | 2 | 0
  Would like - larger screen or font | 4 | 0
  Would like - more rewards | 1 | 0
  Would like - phone version | 1 | 0
  Would like - wider variety of games | 3 | 0
  Would like - nothing, good as is | 14 | 0
  Would like - sound effects | 4 | 0
  Would like - different theme | 4 | 0
  Would like - color blind accessibility | 1 | 0
  Would like - demo video / real human demonstration | 2 | 0
  Would like - personalization | 3 | 0
  Would like - multi-player version | 1 | 0
  Barriers - none | 16 | 0
  Barriers - may be hard for older population to get used to technology | 1 | 0
  Barriers - Setup at home and safety | 3 | 0
  Barriers - learning how to use the app | 1 | 0
  Barriers - equipment (tablet and stand) and equipment setup | 14 | 0
  Barriers - cell phone version would be needed | 1 | 0
  Barriers - cost | 1 | 0
  Barriers - needing family members to help with setup | 1 | 0
  Barriers - adherence to exercises | 1 | 0

14. Primary Outcome: Change in Balance Outcome With the App - Single Leg Balance
Description: The IMU sensor data collected during the exercise performance with and without the Vestibular Rehabilitation App (collected in the same lab visit on the same group of participants) were analyzed to calculate balance measure fluency (a non-dimensional derivative of jerk). This was analyzed to identify differences for the conditions with and without the Vestibular Rehabilitation App
Time Frame: During the testing with the app and during the testing without the app (up to 90 minutes)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Trials With the Vestibular Rehabilitation App | Trials Without the Vestibular Rehabilitation App
Number analyzed (Participants) | 40 | 40
degrees | 0.28 (0.07) | 0.30 (0.07)

ADVERSE EVENTS:
Time Frame: 90 minutes
Arm/Group | Older Adults With Dizziness
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05436067/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05436067/SAP_002.pdf
  • Informed Consent Form (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05436067/ICF_003.pdf